CLINICAL TRIAL: NCT02225249
Title: Examination of the Pulmonary Vascular Barrier in Patients During Lung Transplantation
Brief Title: VASCULUX-examination of the Pulmonary VASCUlar Barrier in Patients During LUng Transplantation
Acronym: VASCULUX
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Dirk Bruegger MD, PD Dr., Ludwig-Maximilians - University of Munich
Other Study IDs: 250-14
Record Dates: First submitted 2014-08-04; First posted 2014-08-26 (Estimated); Last update posted 2014-08-26 (Estimated); Status verified 2014-08

CONDITIONS: End Stage Chronic Obstructive Airways Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood samples will be taken. In summary, 61.2 ml blood will be collected at 7 specific time points.
  Components of the vascular barrier are examined, in detail hyaluronan, syndecan-1, and angiopoietin-2.
Oversight: Data Monitoring Committee: No

SUMMARY:
Lung transplantation is a well established method for surgical therapy for patients with end stage pulmonary disease.

The investigators seek to determine to which extent the pulmonary vascular barrier gets harmed during lung transplantation and whether pulmonary edema after reperfusion can be monitored with measurement of extravascular lung water index (ELWI).

Additionally the investigaors are going to evaluate the correlation between ELWI and shedding of the endothelial glycocalyx.

The study is designed as a prospective observational cohort study.

DETAILED DESCRIPTION:
This study is designed as a single center prospective observational cohort study including only patients who are undergoing lung transplantation due to endstage pulmonary disease.

It is well known that pulmonary edema is one of the major problems following reperfusion of the new organ.

The glycocalyx is located on the apical surface of vascular endothelial cells which line the vascular lumen. The endothelial glycocalyx consists of mainly proteoglycans that covers, among others, leukocyte and thrombocyte receptors and fulfills its principal role in maintaining plasma and vessel wall homeostasis.

In patients undergoing cardiac surgery studies showed regional as well as global ischemia causing an increase of syndecan-1 and heparansulphate in plasma during reperfusion.

The extent of the pulmonary vascular barrier's damage might serve as predictor for postoperative complications as reperfusion edema of the lungs.

To quantify the extent of damage the investigators seek to evaluate the correlation between ELWI and the damage to the vascular barrier. ELWI will be assessed using transpulmonary thermodilution. Components of the vascular barrier will be quantified using ELISA-technique. 10 ml full blood will be drawn at 7 different predifined measurement points named T0-T7 as follows:

* T0 before induction of anesthesia
* T1 before reperfusion of the first lung
* T2 5 min after reperfusion of the first lung
* T3 before reperfusion of the second lung
* T4 5 min after reperfusion of the second lung
* T5 before admission to the intensive care unit
* T6 6h after reperfusion of the last lung
* T7 12h after reperfusion of the last lung

For statistical analysis Student's t-test, Friedman or Wilcoxon rank test will be used, as indicated.

Expected length of the study is 2 years enrolling 30 patients undergoing lung transplantation.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 and younger than 65 years of age
* Scheduled for lung transplantation

Exclusion Criteria:

* Pregnancy
* Necessity of ECMO implementation before induction of general anesthesia
* Mechanical ventilation before lung transplantation

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Eligible for this study are all patients being full of age and younger than 65 years scheduled for lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2014-10; Primary Completion 2016-10 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
Components of the vascular barrier | Repeated mesurements to detect differences from baseline values (T0).
  Repeated measurements of each parameter to detect the difference from baseline values.
  Each component will be measured at time point: T0, T1, T2, T3, T4 and T5.
  Components to be measured [Unit]:
  1. Syndecan-1 [ng/ml]
  2. Hyaluronan [ng/ml]
  3. Heparan-Sulphate [ng/ml]
  4. Angiopoetin-1 [ng/ml]
  5. Angiopoetin-2 [ng/ml]
  Components getting measured using serum or plasma samples.
Extravascular Lung Water Index (ELWI) | repeated measurement of ELWI to detect differences from baseline (T0)
  Increase of the Extravascular Lung Water Index (ELWI) will be determined using thermodilution-method.
  Repeated measurement of ELWI to detect the difference from baseline values.
  Each component will be measured at time point: T0, T5, T6 and T7.
  Unit of measurement: [ml/kg]

SECONDARY OUTCOMES:
Clinical parameters | Repeated measurement of each parameter to detect differences from baseline (T0)
  Follwowing clinicals parameters will be assessed at eacht time point to detect increases or decreases from baseline [Units]:
  Each parameter will be assessed at time point: T0, T1, T2, T3, T4, T5, T6, T7
  1. Oxygenation index [mmHg/FiO2]
  2. Heart rate [beats per min]
  3. Systolic blood pressure [mmHg]
  4. Mean arterial blood pressure [mmHg]
  5. Necessity of extracorporal lung assist [yes/no]
  The investigators assess clinical parameters as oxygenation index, heartrate, blood pressure.

CONTACTS AND LOCATIONS:
Overall Officials: Dirk Bruegger, MD, Principal Investigator — Medical Faculty of Ludwig-Maximilians-University Munich
Locations (1):
- University Hospital of Munich, Munich, Bavaria, Germany